CLINICAL TRIAL: NCT01141218
Title: Survey and Blood Sample Collection for Patients With Lung Cancer Who Never Smoked Cigarettes
Brief Title: Internet-Based Clinical Information and Blood Sample Collection From Patients With Non-Small Cell Lung Cancer Who Never Smoked Cigarettes
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: VICC THO 0938; P30CA068485 (NIH); VU-VICC-THO-0938; IRB# 090568
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Never-smokers with lung cancer
  Interventions: Other: internet-based protocol and physician referral

INTERVENTIONS:
Other: internet-based protocol and physician referral — collection and review, dna and lab biomarker analysis, gene mapping

SUMMARY:
RATIONALE: Gathering health information about patients with non-small cell lung cancer who never smoked cigarettes may help doctors learn more about the disease. Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about cancer and identify biomarkers related to cancer.

PURPOSE: This research study is studying internet-based clinical information and blood sample collection from patients with non-small cell lung cancer who never smoked cigarettes.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the feasibility of an internet-based protocol to collect clinical information and biological specimens from 2,000 never smokers with non-small cell lung cancer.
* To perform genome-wide association studies to identify alleles that predispose to lung cancer in patients that never smoked cigarettes.

OUTLINE:

Patients complete an internet-based questionnaire using the REDCap (Research Electronic Data Capture) survey to determine eligibility. The survey consists of a detailed smoking questionnaire and questions to collect information regarding diagnosis, sex, age, ethnicity, treatment history, and any history of previous malignancies. Blood samples are then collected from eligible patients for DNA and other laboratory analyses. Patients' pathology reports are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* histologically and/or cytologically proven diagnosis of non-small cell lung cancer
* never smoker, defined as having smoked less than 100 cigarettes over one's life-time
* completed survey and inclusion form
* signed informed consent

Exclusion Criteria:

* previous history of cancer (other than lung cancer, except for superficial skin cancers)
* living outside the United States
* patients who cannot read English (as materials will only be written in English)
* unable to understand the protocol or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: never-smokers with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of an internet-based protocol to collect clinical information and biological specimens | Six months following collection of final patient data and biospecimen
Identification of alleles that predispose to lung cancer via genome-wide association studies | one year following collection of final patient data and biospecimen

CONTACTS AND LOCATIONS:
Overall Officials: William Pao, MD, PhD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/